CLINICAL TRIAL: NCT00135616
Title: Randomized Controlled Study Comparing Two Types of Suburethral Slings for the Surgical Treatment of Female Stress Incontinence : TVT and TVT-O.
Brief Title: Treatment of Female Stress Urinary Incontinence: Study Comparing Two Suburethral Slings, Retropubic Approach (TVT) and Trans-Obturator (TVT-O) Approach
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hopital Antoine Beclere (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: xd01
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2007-04-30 (Estimated); Status verified 2007-04

CONDITIONS: Urinary Incontinence, Stress
Keywords: urinary incontinence; stress incontinence; urethra; gynaecologic surgical procedures; suburethral sling
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

INTERVENTIONS:
Device: surgical placement of a suburethral sling tvt or tvt-o

SUMMARY:
The purpose of this study is to compare efficacy and morbidity following the placement of two types of suburethral slings in women presenting with stress urinary incontinence: TVT and TVT-O.

DETAILED DESCRIPTION:
Urinary stress incontinence (USI) is a frequent pathology in women. Surgical treatment is required in 30 to 50% of women presenting with USI. Several surgical techniques are currently available.

At the present time, the placement of suburethral slings is one of the most efficient techniques. Furthermore, the placement of a suburethral sling is known to be associated with a low rate of complications.

Currently, two approaches are available for the placement of a suburethral sling: retropubic approach (TVT) and trans-obturator approach (TVT-O). The efficacy of these two approaches seem equivalents. However, the morbidity related to these two techniques is probably different. In retrospective studies, the retropubic approach is associated with a higher rate of bladder perforation. On the other hand, the trans-obturator approach is supposed to be associated with a higher rate of post-operative pain.

Thus, the purpose of this study is to compare efficacy and morbidity following the placement of two types of suburethral slings in women presenting with stress urinary incontinence: TVT and TVT-O.

ELIGIBILITY:
Inclusion Criteria:

* Woman over 18 years old
* Clinical diagnosis of stress urinary incontinence requiring surgical management
* Must be able to read and sign the consent

Exclusion Criteria:

* Pregnancy
* Anti-coagulant treatment
* Isolated overactive bladder syndrome
* Genital prolapse requiring surgical treatment
* Concomitant hysterectomy

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2005-03; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
pre operative complication: rate of bladder perforation
post operative complication: rate of post-operative pain

SECONDARY OUTCOMES:
efficacy: disparation of urinary incontinence
safety: sexual behaviour

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Deffieux, MD, Principal Investigator — Hopital Antoine Beclere, Clamart, France
Locations (14):
- France (14):
  - CHU Amiens, Amiens
  - Centre Hospitalier Universitaire, Angers
  - CHU Pellegrin, Bordeaux
  - Hopital Saint Andre, Bordeaux
  - CH Chambery, Chambéry
  - Hopital Antoine Beclere, Clamart
  - Hôtel Dieu, Clermont-Ferrand
  - CH Dunkerque, Dunkirk
  - Centre Hospitalier Paul Ardier, Issoire
  - Chu Nancy, Nancy
  - CH Caremeau, Nîmes
  - Hopital Diaconesses Croix Saint Simon, Paris
  - CH Rennes, Rennes
  - CH Rouen, Rouen